CLINICAL TRIAL: NCT06186453
Title: Effectiveness of Bonding-Based Education Intervention for Fathers With Preterm Newborn Infants: Randomised Controlled Study
Brief Title: Effectiveness of Bonding-Based Education Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Uğur Gül, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Akdeniz Nursing Faculty
Record Dates: First submitted 2023-12-16; First posted 2024-01-02 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Preterm; Bonding
Keywords: Father; Bonding; Neonatal Intensive Care Unit
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Father-Preterm Newborn Bonding Program
  Interventions: Behavioral: Father-Preterm Newborn Bonding Program
- Control group (No Intervention): Routine nursing care will be applied

INTERVENTIONS:
Behavioral: Father-Preterm Newborn Bonding Program — B-PreBAP will be applied to the fathers in the intervention group. B-PreBAP application will consist of two stages. The first stage will be passive participation and the second stage will be active participation. B-PreBAP will be applied to fathers for a total of two weeks (Heo & Oh, 2019). In order to prevent interaction between the fathers in the intervention group and the fathers in the control group, the intervention will not be carried out during the routine visiting and information hours of the NICU (13:30-14:30 on Mondays, Wednesdays and Fridays). In the first two interviews, NICU introduction and B-PreBAP education about preterm newborns will be given. In the last three interviews, fathers will be involved in one-to-one practices with their preterm newborns.
  Arms: Intervention group

SUMMARY:
The study aimed to determine the impact of the Father-Preterm Newborn Bonding Programme (B-PreBAP) on fathers' parenting behaviours, stress levels, and support needs. Additionally, the study aimed to investigate the effect of B-PreBAP on the stress levels of preterm newborns.

DETAILED DESCRIPTION:
This study constitutes a part of the doctoral thesis titled "Development of Father-Preterm Newborn Bonding Model".

ELIGIBILITY:
Inclusion Criteria:

1. Characteristics of the father; Turkish speaking Literate 18+ Open to communication and co-operation Fathers who agree to participate in the study will be included
2. Characteristics of the preterm newborn Hospitalised in the NICU from the first postnatal day Preterm newborns born between 32 and 33 weeks

Exclusion Criteria:

1. Characteristics of the father; Has a diagnosed psychiatric diagnosis Having twin preterm newborns
2. Characteristics of the preterm newborn Intubated

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
Father Support Scale: Neonatal Intensive Care Unit | Data will be collected two times as pre-intervention and immediately post-intervention.
  It is a measurement tool to determine the support levels of fathers whose babies are hospitalised in the NICU. As the score on the scale increases, the support needs of fathers whose babies are hospitalized in the neonatal intensive care unit also increase. The total score of the scale is between 0-132 points.

SECONDARY OUTCOMES:
Neonatal Intensive Care Unit Parent Stress Scale | Data will be collected two times as pre-intervention and immediately post-intervention.
  This scale measures the stress levels of parents in NICU. The lowest score is 0 and the highest score is 170. The fathers will be asked about the stress level of each variable in the scale and will be rated from 1 (not stressful) to 5 (extremely stressful). The higher the total score, the higher the stress level.
Postnatal Parental Behaviour Scale | Data will be collected two times as pre-intervention and immediately post-intervention.
  This scale is an observational scale used to measure the behaviour of parents towards their newborn babies. As the total score increases, the interaction between the father and the infant increases. The total score of the scale is between 0-6 points. A higher total score on the scale indicates that the parent has more positive parenting behaviour towards his/her infant.
Neonatal Stress Scale | Data will be collected two times as pre-intervention and immediately post-intervention.
  This scale was developed to measure the stress level of the newborn. As the total score increases, the stress level of the newborn increases. The total score of the scale is between 0-16 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Kepez, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No